CLINICAL TRIAL: NCT00015912
Title: A Phase II Clinical And Biologic Study Of The Combination Of Low Dose Interferon-Alpha And Thalidomide (NSC #66847) For Patients With Relapsed Or Refractory Low-Grade Follicular Lymphoma
Brief Title: Interferon Alfa Plus Thalidomide in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02379; 00-171; CWRU 5Y99; CDR0000068572 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-05-06; First posted 2003-10-15 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Interferon-alpha; Interferon Alfa-n3; Introns; Interferon alpha-2; Thalidomide

ARMS (1):
- Treatment (interferon-alpha, thalidomide) (Experimental): Patients receive interferon alfa subcutaneously every 12 hours and oral thalidomide daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: recombinant interferon alfa; Drug: thalidomide; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: recombinant interferon alfa — Given IV
  Other Names: Alferon N; alpha interferon; IFN-A; Intron A; Roferon-A
Drug: thalidomide — Given orally
  Other Names: Kevadon; Synovir; THAL; Thalomid
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of combining thalidomide with interferon alfa in treating patients who have relapsed or refractory non-Hodgkin's lymphoma. Thalidomide may stop the growth of cancer by stopping blood flow to the tumor. Interferon alfa may interfere with the growth of cancer cells. Combining thalidomide with interferon alfa may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the efficacy of interferon alfa and thalidomide, in terms of response rate, time to progression, and overall survival, in patients with relapsed or refractory low-grade follicular non-Hodgkin's lymphoma.

II. Determine the quantitative and qualitative toxic effects of this regimen in this patient population.

III. Correlate ancillary biological studies with clinical endpoints in these patients treated with this regimen.

OUTLINE:

Patients receive interferon alfa subcutaneously every 12 hours and oral thalidomide daily in the absence of disease progression or unacceptable toxicity. Patients are followed every 6 months until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed relapsed or refractory low-grade follicular non-Hodgkin's lymphoma (NHL)

  * WHO grade 1 or 2
  * Failure to achieve a complete or partial remission after prior treatment regimen
  * Relapse or disease progression within 30 days after prior treatment regimen
* No histologic transformation to aggressive NHL or areas of diffuse NHL
* At least 1 measurable lesion by CT scan, MRI, or chest x-ray
* Tissue in the form of tissue blocks available
* No brain metastasis or primary brain tumors
* Performance status - ECOG 0-1
* More than 3 months
* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 8.5 g/dL
* Bilirubin no greater than 1.5 mg/dL
* SGOT/SGPT no greater than 2.5 times upper limit of normal
* PT (or INR)/PTT normal or not clinically significant
* No preexisting liver disease
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance greater than 60 mL/min
* No uncompensated coronary artery disease
* No myocardial infarction or severe/unstable angina within the past 6 months
* No active infection
* No prior gastrointestinal disorder that would interfere with thalidomide absorption
* No preexisting autoimmune disease
* No medical, psychological, or social problem that would preclude study participation
* No uncontrolled or untreated depression
* No emotional disorder or substance abuse
* No prior seizures or potential risk factors for development of seizures
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test at baseline, weekly for 4 weeks, and then every 2-4 weeks thereafter while on study
* Fertile female patients must use 1 highly active method and 1 additional effective method of contraception for 4 weeks before, during, and for 4 weeks after study
* Fertile male patients must use effective barrier contraception during and for 4 weeks after study participation
* No more than 1 prior course of unconjugated monoclonal antibody therapy
* No prior conjugated monoclonal antibody (radiolabeled or immunotoxin) therapy
* No prior interferon alfa
* No concurrent hematopoietic growth factors or other cytokines
* No concurrent monoclonal antibodies
* No more than 2 prior chemotherapy regimens (single agent or combination)
* At least 28 days since prior chemotherapy
* No concurrent chemotherapy
* At least 28 days since prior corticosteroid therapy
* Prior or concurrent megestrol allowed
* No concurrent corticosteroids
* No concurrent hormonal therapy
* Prior palliative radiotherapy to nontarget lesions allowed
* No prior radiotherapy to all sites of measurable disease
* No prior extensive radiotherapy to more than 20% of bone marrow
* No concurrent palliative radiotherapy
* At least 14 days since prior major surgery
* No prior major upper gastrointestinal surgery
* No other concurrent cytotoxic agents
* No other concurrent investigational therapy
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2001-07; Primary Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Response rate (complete and partial) | Up to 2 years

SECONDARY OUTCOMES:
Time to progression | Up to 2 years
  Kaplan-Meier estimates will be determined.
Overall survival | Up to 2 years
  Kaplan-Meier estimates will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: John Sweetenham, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Colorado, United States